CLINICAL TRIAL: NCT03174483
Title: Effects of Hypertonic Saline and Fluticasone Nasal Sprays on Radiologic Scoring of Patients With Chronic Sinusitis and Nasal Polyps
Brief Title: Radiologic Scoring of Patients With Chronic Sinusitis and Nasal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Abdel aal Mekhamar Abdel aal, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSCS
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypertonic saline (Experimental): nasal spray will be used twice daily
  Interventions: Drug: Hypertonic saline
- fluticasone (Active Comparator): nasal spray will be used once daily
  Interventions: Drug: Fluticasone Nasal

INTERVENTIONS:
Drug: Hypertonic saline — nasal spray
  Arms: hypertonic saline
Drug: Fluticasone Nasal — nasal spray
  Arms: fluticasone

SUMMARY:
To detect the effect of hypertonic saline and fluticasone sprays on computed tomography scan of paranasal sinuses of patients having chronic sinusitis and/or nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic sinusitis and/or nasal polyps.

Exclusion Criteria:

* Patients with previous nasal or sinus surgery.
* Patients with sinonasal Malignancy.
* Immunocompromised patients.
* Patients with ciliary motility disorders.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of patient with normal radiological scoring | 1 month
  the score used is Lund Mackay radiological scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No